CLINICAL TRIAL: NCT07094971
Title: Safety and Efficacy of Pure Impact to Strengthen and Tone Abdomen, Quadriceps and Glutes Muscles
Brief Title: Pure Impact Treatment to Strengthen and Tone Abdomen, Quadriceps and Glutes Muscles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sofwave27
Record Dates: First submitted 2025-07-29; First posted 2025-07-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Muscle Tone; Muscle Strength
Keywords: Abdomen; Hamstring; Quadriceps; Glutes; skin laxity; muscle tone; muscle strength; muscle firm
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Muscle strength (Experimental): Pure Impact is an EMS module. Pure Impact generates electrical impulses, which are delivered through electrodes on the skin in direct proximity to the muscles to be stimulated.
  Interventions: Device: Pure Impact
- Control (No Intervention): Control group will be followed but will not be treated.

INTERVENTIONS:
Device: Pure Impact — Pure Impact is an EMS module. Pure Impact generates electrical impulses, which are delivered through electrodes on the skin in direct proximity to the muscles to be stimulated.
  Arms: Muscle strength

SUMMARY:
Open-label, non-randomized, prospective, single-center, self-controlled clinical study.

DETAILED DESCRIPTION:
Eligible subjects will be divided into two groups. The test group will include 15-22 subjects who will be treated to revive their body's functional potential, and the control group will include 15-22 subjects, who will not be treated.

The Test group will arrive to 6 Pure Impact sessions and to 4 weeks follow-up visit; while the control group will arrive to 3 visits, which are equivalent to before first treatment, last treatment (5 weeks after first visit) and 4 weeks after the second visit (equivalent to 4 weeks follow-up visit of the test group).

Subjects of the test group will receive 6 Pure Impact treatments on the abdomen and quadriceps, and/or hamstring and glutes once a week.

First treatment may be administered after the enrolment and screening at the first visit, or it may occur later following the enrolment and screening activities based on site scheduling availabilities.

Overall, all treatments are done within 6 weeks.

All subjects will return to the clinic for follow-up visit at 4±1 weeks post last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 25 years of age and ≤ 60 years of age.
2. Not pregnant or lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide) or abstinence.
3. Desire to undergo treatments on abdomen and quadriceps and/or on hamstring and glutes for strength and tone muscles.
4. Subject agrees to maintain their weight within 5% of total body weight and avoid significant dietary or exercise changes during the study.
5. Able and willing to comply with all visits, treatments and evaluations schedules and requirements.
6. Willing to have research photos taken of treatment areas.
7. Able to understand and provide written Informed Consent.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
2. Medical disorder that would hinder the wound healing or immune response (such as blood disorder) including but not limited to arterial circulation disorders in lower limbs, inflammatory disease, etc.
3. Active malignancy or history of malignancy in the past 5 years.
4. Suffering from significant concurrent illness, such as cardiac disorders, sensory disturbances, diabetes (type I or II), epilepsy, lupus, porphyria, pertinent neurological disorders, uncontrolled hypertension, or liver or kidney disease (i.e. any disease state that in the opinion of the investigator may interfere with the anesthesia, treatment, or healing process).
5. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
6. BMI < 18 or >35kg/m2
7. Non-stable weight nominally ±5% in the past month.
8. Active implanted device such as a pacemaker, defibrillator, drug delivery system or any other metallic or electric implant anywhere in the body.
9. Permanent implant in the treated area such as metal plates, screws and metal piercing, silicone implants or an injected chemical substance, unless deep enough in the periosteal plane.
10. History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.) at the last 2 years.
11. History of prior surgery in the treated areas at the last 2 years.
12. Excessive subcutaneous fat on the treated areas.
13. Abdominal or inguinal hernia
14. Any active condition in the treatment area, such as open wounds, sores, psoriasis, eczema, and rash.
15. Any sensitivity for hydrogel (Pure Impact electrodes pads are made of hydrogel).
16. History of chronic drug or alcohol abuse.
17. Muscle atrophy.
18. Need for muscle rehabilitation.
19. Persistent pain at the treated area.
20. Inability to understand the protocol or to give informed consent.
21. Unable or unwilling to comply with the study requirements and procedures.
22. Currently enrolled in a clinical study of any other unapproved investigational drug or device.
23. Any other condition that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.
24. Presence of any active systemic or local infections.
25. Significant scarring in the area to receive study treatment.
26. Suspected or diagnosed heart problems.
27. Areas of the skin that lack normal sensation.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Improvement rate of the muscles strength | 1 Month post last treatment follow up visit
  Higher improvement rate of the muscles strength tests at the test group compared to the control group using series of exercises tests including questionnaire, and a functional evaluation of the muscles of the abdomen, quadriceps, and glutes.

CONTACTS AND LOCATIONS:
Overall Officials: Ahlam Safadi, BSC, Study Director — Sofwave Medical LTD
Locations (1):
- Movassaghi Plastic Surgery & Ziba Medical Spa, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No